CLINICAL TRIAL: NCT06372483
Title: A Randomised, Double-Blind, Placebo-Controlled, Single Dose Trial Evaluating Different Doses of Intravenously Administered VMX-C001 and to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of VMX-C001 in Healthy Subjects (Part 1) and in Combination with a Selected FXa Direct Oral Anticoagulant (DOAC) in Healthy Older Subjects (Part 2)
Brief Title: Single Dose Trial of VMX-C001 in Healthy Subjects with and Without FXa Direct Oral Anticoagulant
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VarmX B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMX-C001-03; 2023-507059-32-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-15; First posted 2024-04-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders | interventions — Rivaroxaban; apixaban; Tablets; edoxaban

STUDY DESIGN:
Intervention Model Description: Placebo controlled, single dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Part 1, Cohort 1:1 - VMX-C001 (Experimental): Single dose active.
  Interventions: Drug: VMX-C001
- Part 1, Cohort 1:1 - Placebo (Placebo Comparator): Single dose placebo.
  Interventions: Drug: Placebo
- Part 2, Cohort 2:1 - VMX-C001 + Rivaroxaban (Experimental): Single dose active in combination with DOAC.
  Interventions: Drug: VMX-C001; Drug: Rivaroxaban 20 mg Oral Tablet
- Part 2, Cohort 2:1 - Placebo + Rivaroxaban (Placebo Comparator): Single dose placebo in combination with DOAC.
  Interventions: Drug: Placebo; Drug: Rivaroxaban 20 mg Oral Tablet
- Part 2, Cohort 2:2 - VMX-C001 + DOAC (Experimental): Optional cohort - Single dose active in combination with selected DOAC.
  Interventions: Drug: VMX-C001; Drug: Rivaroxaban 20 mg Oral Tablet; Drug: Apixaban 5 mg Oral Tablet; Drug: Edoxaban 60 mg Oral Tablet
- Part 2, Cohort 2:2 - Placebo + DOAC (Placebo Comparator): Optional cohort - Single dose placebo in combination with selected DOAC.
  Interventions: Drug: Placebo; Drug: Rivaroxaban 20 mg Oral Tablet; Drug: Apixaban 5 mg Oral Tablet; Drug: Edoxaban 60 mg Oral Tablet
- Part 2, Cohort 2:3 - VMX-C001 + DOAC (Experimental): Optional cohort - Single dose active in combination with selected DOAC.
  Interventions: Drug: VMX-C001; Drug: Rivaroxaban 20 mg Oral Tablet; Drug: Apixaban 5 mg Oral Tablet; Drug: Edoxaban 60 mg Oral Tablet
- Part 2, Cohort 2:3 - Placebo + DOAC (Placebo Comparator): Optional cohort - Single dose placebo in combination with selected DOAC.
  Interventions: Drug: Placebo; Drug: Rivaroxaban 20 mg Oral Tablet; Drug: Apixaban 5 mg Oral Tablet; Drug: Edoxaban 60 mg Oral Tablet
- Part 2, Cohort 2:4 - VMX-C001 + DOAC (Experimental): Optional cohort - Single dose active in combination with selected DOAC.
  Interventions: Drug: VMX-C001; Drug: Rivaroxaban 20 mg Oral Tablet; Drug: Apixaban 5 mg Oral Tablet; Drug: Edoxaban 60 mg Oral Tablet
- Part 2, Cohort 2:4 - Placebo + DOAC (Placebo Comparator): Optional cohort - Single dose placebo in combination with selected DOAC.
  Interventions: Drug: Placebo; Drug: Rivaroxaban 20 mg Oral Tablet; Drug: Apixaban 5 mg Oral Tablet; Drug: Edoxaban 60 mg Oral Tablet

INTERVENTIONS:
Drug: VMX-C001 — VMX-C001 is human factor X engineered to be insensitive to factor Xa DOACs
  Arms: Part 1, Cohort 1:1 - VMX-C001; Part 2, Cohort 2:1 - VMX-C001 + Rivaroxaban; Part 2, Cohort 2:2 - VMX-C001 + DOAC; Part 2, Cohort 2:3 - VMX-C001 + DOAC; Part 2, Cohort 2:4 - VMX-C001 + DOAC
Drug: Placebo — VMX-C001 matched placebo
  Arms: Part 1, Cohort 1:1 - Placebo; Part 2, Cohort 2:1 - Placebo + Rivaroxaban; Part 2, Cohort 2:2 - Placebo + DOAC; Part 2, Cohort 2:3 - Placebo + DOAC; Part 2, Cohort 2:4 - Placebo + DOAC
Drug: Rivaroxaban 20 mg Oral Tablet — Fxa DOAC
  Arms: Part 2, Cohort 2:1 - Placebo + Rivaroxaban; Part 2, Cohort 2:1 - VMX-C001 + Rivaroxaban; Part 2, Cohort 2:2 - Placebo + DOAC; Part 2, Cohort 2:2 - VMX-C001 + DOAC; Part 2, Cohort 2:3 - Placebo + DOAC; Part 2, Cohort 2:3 - VMX-C001 + DOAC; Part 2, Cohort 2:4 - Placebo + DOAC; Part 2, Cohort 2:4 - VMX-C001 + DOAC
Drug: Apixaban 5 mg Oral Tablet — Fxa DOAC
  Arms: Part 2, Cohort 2:2 - Placebo + DOAC; Part 2, Cohort 2:2 - VMX-C001 + DOAC; Part 2, Cohort 2:3 - Placebo + DOAC; Part 2, Cohort 2:3 - VMX-C001 + DOAC; Part 2, Cohort 2:4 - Placebo + DOAC; Part 2, Cohort 2:4 - VMX-C001 + DOAC
Drug: Edoxaban 60 mg Oral Tablet — Fxa DOAC
  Arms: Part 2, Cohort 2:2 - Placebo + DOAC; Part 2, Cohort 2:2 - VMX-C001 + DOAC; Part 2, Cohort 2:3 - Placebo + DOAC; Part 2, Cohort 2:3 - VMX-C001 + DOAC; Part 2, Cohort 2:4 - Placebo + DOAC; Part 2, Cohort 2:4 - VMX-C001 + DOAC

SUMMARY:
A single centre, double-blind, randomized, placebo-controlled single dose study to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of VMX-C001, conducted in two parts:

Part 1: Single dose of VMX-C001 or placebo in healthy volunteers.

Part 2: Single dose of VMX-C001 or placebo in combination with a selected factor 10a (FXa) direct oral anticoagulant (DOAC) in healthy older subjects.

ELIGIBILITY:
Inclusion Criteria:

1. In Part 1, men and women of any ethnic origin between 18 and 49 years of age, in Part 2, men and women of any ethnic origin between 50 and 79 years of age, inclusive, at the time of Screening.
2. Male subjects must be willing to use appropriate contraception, such as a condom, and to refrain from sperm donation during the study and until 90 days after study drug administration.
3. Women of child-bearing potential must agree not to attempt to become pregnant and to use a highly effective form of birth control during the study and for 90 days after study drug administration when their sexual partner has not been vasectomized. Highly effective forms of birth control entail the use of combined (estrogen- and progestogen-containing) or progestogen-only hormonal contraception associated with inhibition of ovulation, an intrauterine device (IUD), an intrauterine hormone-releasing system (IUS) or abstinence.
4. Postmenopausal women must have had ≥12 months of spontaneous amenorrhea (with documented follicle-stimulating hormone (FSH) >33.4 IU/L).
5. Surgically sterile women are defined as those who have had a surgical bilateral oophorectomy with or without hysterectomy, total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, the reproductive status of the woman has to be confirmed by follow-up hormone level assessment. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.
6. Subject must weigh between 60 and 120 kg, inclusive, and must have a BMI between 18.0 and 30.0 kg/m2, inclusive, at Screening and on Day -1.
7. Subject must be in good health, as determined by a medical history, physical examination, 12-lead ECG, and clinical laboratory evaluations (congenital non hemolytic hyperbilirubinemia is acceptable).
8. Subject is willing and able to give their written informed consent to participate in the study and to abide by the study restrictions.
9. Subject has good upper limb venous access.

Exclusion Criteria:

1. The subject has taken tenoxicam in the 35 days prior to the first administration of study drug or FXa DOAC or has taken piroxicam in the two weeks prior to the first administration of study drug or FXa DOAC.
2. The subject has taken any non-aspirin, non-piroxicam, non-steroidal anti-inflammatory drug (NSAID) in the week prior to the first administration of study drug or FXa DOAC.
3. The subject requires or has taken during the month prior to first administration of study drug or FXa DOAC, vitamin K for therapeutic reasons. Vitamin K not taken for therapeutic purposes is acceptable, e.g., as part of a multivitamin supplement.
4. The subject is receiving or requires, for any cause, any anticoagulant or antiplatelet therapy including warfarin, clopidogrel or aspirin or any other anticoagulant or antiplatelet agent or has used these therapies in the month prior to the first administration of study drug or FXa DOAC.
5. The subject has received any prescribed oral, systemic or topical medication, including any vaccinations, within 14 days prior to the first administration of study drug or FXa DOAC (with the exception of contraceptives), unless in the opinion of the Principal Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
6. The subject has used any non-prescribed systemic or topical medication (including herbal remedies) within one week prior to the first administration of study drug or FXa DOAC (with the exception of oral vitamin/mineral supplements [including those that contain vitamin K when not taken for therapeutic purposes] and paracetamol), unless in the opinion of the Principal Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
7. The subject is currently participating in a clinical study, e.g. attending follow-up visits or has been administered an investigational drug (new chemical or biological entity) within 1 month (for small molecules) or 3 months (for biologicals) prior to administration of the study drug.
8. The subject has donated ≥500 mL blood, plasma, or platelets in the 3 months prior to Screening or any other blood amount within 30 days prior to Screening.
9. Because of an increased risk of thrombosis subjects with known diabetes mellitus or a fasted glucose ≥7.0 mmol/L at Screening.
10. The subject has any bleeding diathesis, any increased risk of bleeding or, in the opinion of the Principal Investigator, is at increased risk of the consequences of bleeding including but not limited to the following:

    1. gastro-intestinal ulceration within the last 3 months;
    2. known or suspected oesophageal varices;
    3. vascular aneurysms or known arteriovenous malformations;
    4. history of known major intraspinal or intracerebral vascular abnormalities;
    5. history of brain, spinal or ophthalmic surgery within the last year;
    6. any intracranial hemorrhage;
    7. uncontrolled severe hypertension.
11. The subject has, in the opinion of the Principal Investigator, any increased risk of thrombosis or thromboembolism including any known thrombophilia, such as antiphospholipid syndrome, or any past history of provoked or unprovoked arterial or venous thrombosis, including thromboembolism.
12. The subject has a significant history of drug allergy, as determined by the Principal Investigator.
13. The subject has at Screening or on Day -1, a supine blood pressure or supine pulse rate ≥ 150/95 mmHg and >100 beats per minute (bpm), respectively, or < 90/40 mmHg and 40 bpm, respectively, confirmed by a repeat assessment.
14. For Part 1, the subject consumes >21 alcoholic drinks/week for men or >14 alcoholic drinks/week for women (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1 measure [25 mL] of spirits) or has a significant history of alcoholism or drug/chemical abuse, as determined by the Principal Investigator. For Part 2, the subject consumes >14 alcoholic drinks/week or has a significant history of alcoholism or drug/chemical abuse, as determined by the Principal Investigator.
15. The subject has a positive drug screen, alcohol test or cotinine test result at Screening or on Day -1, confirmed by repeat testing.
16. The female subject has a positive pregnancy test at Screening or on Day -1 or is lactating.
17. The subject currently smokes or uses nicotine-containing products. Former smokers will be eligible, provided they have not smoked for at least 1 month prior to administration of the study drug.
18. The subject has, or has a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, hematological, or other major disorders, as determined by the Principal Investigator.
19. The subject has a positive Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody test result at Screening.
20. The subject has an abnormality in the 12-lead ECG at Screening or on Day -1 that, in the judgement of the Principal Investigator may, during the study, interfere with the interpretation of 12-lead ECG results, including average QTcF interval >450 msec for men or >470 msec for women, 2nd or 3rd degree atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolff-Parkinson-White Syndrome, defined as average PR<110 msec, confirmed by a triplicate repeat ECG.
21. The subject has any other condition that, in the opinion of the Principal Investigator, would compromise the safety of the subject or the subject's ability to comply with the protocol and complete the study.
22. The subject has renal insufficiency (serum creatinine level > 1.25 times upper limit of normal (ULN) or estimated glomerular filtration rate (eGFR) of <60 mL/min*1.73m2).
23. The subject has active liver disease (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >1.5x ULN, or total bilirubin > 1.5x ULN at Screening or on Day -1. One re-test is allowed).
24. The subject has previously participated in a clinical study with VMX-C001.

    Additional exclusion criteria for Part 2 only:
25. Because of an effect on FXa DOACs, subjects are to be excluded if he/she receives or has received medication that is an inhibitor of P-glycoprotein or CYP3A4. (e.g., clarithromycin, erythromycin and azole-antimycotics such as ketoconazole, itraconazole, voriconazole and osaconazole or HIV protease inhibitors.) within 30 days prior to first administration of FXa DOAC.
26. Because of an effect on FXa DOACs, subjects are to be excluded if he/she receives or has received treatment with CYP3A4 inducers (e.g., St. John's wort, rifampicin, phenytoin, carbamazepine, phenobarbital) within 30 days prior to first administration of FXa DOAC.
27. Because of an effect on FXa DOACs, subjects are to be excluded if he/she receives or has received treatment with selective serotonin reuptake inhibitors (SSRIs) or selective noradrenaline reuptake inhibitors (SNRIs) within 30 days prior to first administration of FXa DOAC.
28. The subject has any contra-indication to treatment with FXa DOACs.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] (Part 1) | From dosing up to Day 28
  Number of Subjects with One of More Drug Related Adverse Events (AEs) or any Serious AEs
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] (Part 2) | From dosing up to Day 31
  Number of Subjects with One of More Drug Related Adverse Events (AEs) or any Serious AEs
PK of VMX-C001 in plasma - Cmax | Up to 7 days post VMX-C001 dose
  Maximal concentration in plasma
PK of VMX-C001 in plasma - tmax | Up to 7 days post VMX-C001 dose
  Time of maximal concentration in plasma
PK of VMX-C001 in plasma - t1/2 | Up to 7 days post VMX-C001dose
  Terminal elimination half-life in plasma
PK of VMX-C001 in plasma - AUC0-last | Up to 7 days post VMX-C001 dose
  Area under the concentration-time curve from time of dosing to last measurable concentration in plasma
PK of VMX-C001 in plasma - AUC0-inf | Up to 7 days post VMX-C001 dose
  Area under the concentration-time curve from time of dosing extrapolated to infinity in plasma
PK of VMX-C001 in plasma - Lambda z | Up to 7 days post VMX-C001 dose
  Terminal elimination rate constant
PK of VMX-C001 in plasma - CL | Up to 7 days post VMX-C001 dose
  Total body clearance
PK of VMX-C001 in plasma - Vz | Up to 7 days post VMX-C001 dose
  Apparent volume of distribution
DOAC plasma concentrations (Part 2) | Up to Day 10
Change in Prothrombin time (PT) following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
Change in activated partial thromboplastin time (aPTT) following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
Change in D-dimer following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
Change in prothrombin fragments F1 and 2 following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
  Mean and median values, subjects on active treatment per group versus placebo
Change in thrombin generation, measured by lag time, following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
  Mean and median values, subjects on active treatment per group versus placebo
Change in thrombin generation, measured by endogenous thrombin potential, following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
  Mean and median values, subjects on active treatment per group versus placebo
Change in thrombin generation, measured by peak height, following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
  Mean and median values, subjects on active treatment per group versus placebo
Change in thrombin generation, measured by time to peak, following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
  Mean and median values, subjects on active treatment per group versus placebo
Change in thrombin generation, measured by velocity index, following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
  Mean and median values, subjects on active treatment per group versus placebo
Change in thrombin generation, measured by time to tail, following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
  Mean and median values, subjects on active treatment per group versus placebo
Change in diluted prothrombin time (dPT) following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
Change in diluted Russell Viper Venom time (dRVVT) following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose
Change in real time activated clotting time (ACT) following dosing with VMX-C001 | Up to 7 days post VMX-C001 dose

SECONDARY OUTCOMES:
Antibodies against VMX-C001 in plasma | Up to 28 days post VMX-C001 dose
  Percentage of patients positive (active vs placebo), and titer (percentage of patients tested positive for each titer measured)
Antibodies against human coagulation FX in plasma | Up to 28 days post VMX-C001 dose
  Percentage of patients positive (active vs placebo), and titer (percentage of patients tested positive for each titer measured)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands